CLINICAL TRIAL: NCT03656822
Title: Data Visualization of Kidney and Prostate Tumors Using Routine Pre-Operative Imaging, 3D Printed, and 3D Virtual Reality Models
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-00697
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Routine imaging such as CT or MRI: Subjects will undergo routine pre-operative imaging and will be randomized into 3 groups for data visualization. This group will receive data visualization using routine clinical imaging,
  Interventions: Diagnostic Test: Routine CT; Diagnostic Test: Routine MRI
- Routine imaging (CT or MRI) with a 3D printed model: Subjects will undergo routine pre-operative imaging and will be randomized into 3 groups for data visualization. This group will receive data visualization using routine clinical imaging with a 3D printed anatomical mode
  Interventions: Diagnostic Test: Routine imaging CT with a 3D printed model; Diagnostic Test: Routine imaging MRI with a 3D printed model
- Routine imaging (CT or MRI) with a VR model: Subjects will undergo routine pre-operative imaging and will be randomized into 3 groups for data visualization. This group will receive data visualization using routine clinical imaging with a 3D VR anatomical model
  Interventions: Diagnostic Test: Routine imaging CT with a VR model; Diagnostic Test: Routine imaging MRI with a VR model

INTERVENTIONS:
Diagnostic Test: Routine CT — CAT (Computerized Axial Tomography) scan, is a noninvasive X-ray test that is used to diagnose a variety of medical conditions.
  Groups: Routine imaging such as CT or MRI
Diagnostic Test: Routine imaging CT with a 3D printed model — CAT (Computerized Axial Tomography) scan, is a noninvasive X-ray test that is used to diagnose a variety of medical conditions + 3D Printed Model
  Groups: Routine imaging (CT or MRI) with a 3D printed model
Diagnostic Test: Routine imaging MRI with a 3D printed model — will measure post-operative lesion volume as visualized on the post-operative MRI + 3D Printed Model
  Groups: Routine imaging (CT or MRI) with a 3D printed model
Diagnostic Test: Routine MRI — will measure post-operative lesion volume as visualized on the post-operative MRI
  Groups: Routine imaging such as CT or MRI
Diagnostic Test: Routine imaging CT with a VR model — CAT (Computerized Axial Tomography) scan, is a noninvasive X-ray test that is used to diagnose a variety of medical conditions + VR Model
  Groups: Routine imaging (CT or MRI) with a VR model
Diagnostic Test: Routine imaging MRI with a VR model — will measure post-operative lesion volume as visualized on the post-operative MRI + VR Model
  Groups: Routine imaging (CT or MRI) with a VR model

SUMMARY:
The purpose of this study is to determine whether adding new methods of data visualization to routine clinical care will improve (i) surgical planning and (ii) surgical outcomes in patients with kidney and prostate tumors.

DETAILED DESCRIPTION:
This early phase I trial studies how well indwelling pleural catheters with doxycycline work compared to indwelling pleural catheters alone in treating participants with malignant pleural effusions. These types of catheters are commonly used to treat pleural effusions (build-up of fluid in the lungs). Doxycycline is an antibiotic that is also used to treat pleural effusions. It is not yet known whether giving doxycycline with indwelling pleural catheters works better than indwelling pleural catheters alone in treating participants with cancerous pleural effusions.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with MPE undergoing IPC placement
* Sufficient mental capacity to provide informed consent and answer Short-Form Six-Dimension health index (SF-6D) and Borg score questions

Exclusion Criteria:

* Patients undergoing pleurodesis for benign disease (e.g., spontaneous pneumothorax)
* Inability or unwillingness to give informed consent
* Inability to perform phone call and clinical follow-up at MD Anderson Cancer Center (MDACC)
* Pregnancy
* Previous intrapleural therapy for MPE on the same side
* Eastern Cooperative Oncology Group (ECOG) of 4 and life expectancy ≤ 2 weeks
* Doxycycline allergy
* Extensive loculations or hydropneumothorax or other contraindication to pleurodesis
* Chylous effusions associated with malignant disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have scheduled to have kidney or prostate cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Measure of Operative Time | Post Surgery
  measure of the amount of time it takes surgeon to remove tumor

CONTACTS AND LOCATIONS:
Overall Officials: Hersh Chandarana, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States